CLINICAL TRIAL: NCT02854995
Title: Circumcision Versus Preputioplasty for BXO in Children: A Feasibility Randomised Controlled Trial
Brief Title: Circumcision Versus Preputioplasty for BXO in Children
Acronym: BXO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alder Hey Children's NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BXO
Record Dates: First submitted 2016-07-22; First posted 2016-08-04 (Estimated); Last update posted 2018-11-09 (Actual); Status verified 2017-10

CONDITIONS: Balanitis Xerotica Obliterans (BXO)
MeSH Terms: conditions — Balanitis Xerotica Obliterans | interventions — Circumcision, Male

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- circumcision (Other): (i) circumcision: this will be a standard surgical circumcision whereby the prepuce (foreskin of the penis) is excised and the cut edge of the outer prepuce sutured to the cut edge of the inner prepuce.
  Interventions: Procedure: circumcision
- preputioplasty with intralesional injection of triamcinolone (Other): (ii) preputioplasty with intralesional injection of triamcinolone: longitudinal incisions will be placed in the area of phimosis, and these will be sutured transversely to allow the prepuce to become retractile.
  Interventions: Procedure: preputioplasty with intralesional injection of triamcinolone:

INTERVENTIONS:
Procedure: circumcision — (i) circumcision: this will be a standard surgical circumcision whereby the prepuce (foreskin of the penis) is excised and the cut edge of the outer prepuce sutured to the cut edge of the inner prepuce. The two study team members performing the surgery in this trial (HC and SK) will be free to choose the method of circumcision (e.g. guillotine vs. sleeve) as this is not thought to influence outcome. The foreskin will be sent for histological analysis.
  Arms: circumcision
Procedure: preputioplasty with intralesional injection of triamcinolone: — (ii) preputioplasty with intralesional injection of triamcinolone: this will be performed as described by Wilkinson et al.[5] Briefly, longitudinal incisions will be placed in the area of phimosis, and these will be sutured transversely to allow the prepuce to become retractile. A biopsy of an area of affected foreskin will be sent for histological analysis. The intention will be to perform three incisions (tri-radiate) but the final decision on how many will be made by the operating surgeon and based on the appearance of the prepuce and result of initial incision(s). Once the prepuce is felt to be freely retractile, 1 - 3 mL of triamcinolone (Adcortyl Bristol-Myers Squibb 10 mg/mL) will be injected intradermally around the circumference of the affected foreskin using a 25-gauge needle.
  Arms: preputioplasty with intralesional injection of triamcinolone

SUMMARY:
Traditionally, BXO is managed with circumcision (surgical removal of the foreskin) and this approach has long been held as the 'gold standard. Whilst this may be curative in many cases, it has been shown that 20% of boys require a further operative procedure on their penis to widen the urethral opening (to treat meatal stenosis)

An alternative to circumcision was proposed: a preputioplasty (surgery to widen the opening of the foreskin) was combined with injection of steroids into the affected foreskin. Subsequently, the same group compared the outcomes of this technique with circumcision, and reported circumcision was successfully avoided in 92% of the preputioplasty group. In addition, the rate of meatal stenosis (narrowing of the urethral opening requiring surgery) was significantly lower (6% vs 19%, P = .034 ). Preputioplasty may therefore: (i) offer protection against meatal stenosis and reduce the requirement for further surgery; and (ii) offer the benefit of retaining the foreskin, the function of which, while debated, likely includes sexual function. In view of these potential benefits, authors have called for a randomised trial to compare circumcision to preputioplasty and injection of steroids.

DETAILED DESCRIPTION:
The interventions to be compared are operations to treat BXO called:

(i) circumcision: this will be a standard surgical circumcision whereby the prepuce (foreskin of the penis) is excised and the cut edge of the outer prepuce sutured to the cut edge of the inner prepuce. The two study team members performing the surgery in this trial (HC and SK) will be free to choose the method of circumcision (e.g. guillotine vs. sleeve) as this is not thought to influence outcome. The foreskin will be sent for histological analysis.

(ii) preputioplasty with intralesional injection of triamcinolone. Briefly, longitudinal incisions will be placed in the area of phimosis, and these will be sutured transversely to allow the prepuce to become retractile. A biopsy of an area of affected foreskin will be sent for histological analysis. The intention will be to perform three incisions (tri-radiate) but the final decision on how many will be made by the operating surgeon and based on the appearance of the prepuce and result of initial incision(s). Once the prepuce is felt to be freely retractile, 1 - 3 mL of triamcinolone (Adcortyl Bristol-Myers Squibb 10 mg/mL) will be injected intradermally around the circumference of the affected foreskin using a 25-gauge needle.

These procedures are established treatments for BXO and currently in use by the trial surgeons in the same setting as the trial.The preputioplasty with injection of triamcinolone procedure has previously been approved by the Alder Hey Children's Hospital NHS Trust Clinical Development Evaluation Group (CDEG).

ELIGIBILITY:
Inclusion Criteria:

* aged between 2 and 16 years
* diagnosed with BXO
* require surgery to treat BXO

Exclusion Criteria:

* previous penile surgery
* circumcision or preputioplasty medically contraindicated

Ages: 2 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2018-01-31 (Actual); Study Completion 2018-11-07 (Actual)

PRIMARY OUTCOMES:
Recruitment Rate | 12 months
  Recruitment Rate including reasons for non-recruitment.
Protocol Adherence | 12 months
  Rate of adherence to protocol-data collected by study team
Drop Out | 12 months
  Rate of drop-out from the study

SECONDARY OUTCOMES:
Patient Satisfaction | 6 weeks, 3 months and 12 months
  Satisfaction with treatment process (at 6 weeks) and overall outcome (3 and 12 months) - data collected by questionnaire
Clinical outcomes-Readmissions to hospital | 30 days
  Readmissions to hospital (number of readmissions within 30 days)
Clinical outcomes-Surgical complications | 72 hours
  Surgical complications: specifically, wound infection (defined by intention to treat with antibiotics); urinary retention requiring intervention; post-operative bleeding requiring return to theatre
Clinical outcomes-Return to theatre | 30 days
  Return to theatre for a complication (within 30 days)
Clinical outcomes-patient satisfaction | 3 months & 1 year
  Medium term patient satisfaction (questionnaire at 3 months and 1 year)
Clinical outcomes-functional outcomes | 6 weeks, 3 months & 1 year
  Functional outcomes: urinary flow rate at 6 weeks, 3 months and 1 year
Clinical outcomes-Subsequent penile surgery | 1 year
  Subsequent penile surgery (other than for early complication): e.g. meatal procedure, re-do preputioplasty or circumcision

CONTACTS AND LOCATIONS:
Locations (1):
- Alder Hey Children's Hospital, Liverpool, Merseyside, United Kingdom

REFERENCES:
- [Derived] Lansdale N, Arthur F, Corbett HJ. Circumcision versus preputioplasty for balanitis xerotica obliterans: a randomised controlled feasibility trial. BJU Int. 2021 Dec;128(6):759-765. doi: 10.1111/bju.15508. Epub 2021 Jul 11. PMID 34110689